CLINICAL TRIAL: NCT05012787
Title: A Double-Blind, Randomized, Controlled, Phase 3 Study to Evaluate the Safety and Immunogenicity of CpG 1018/Alum-adjuvanted SCB-2019 in Individuals Aged 18 and Above With Chronic Immune-Mediated Inflammatory Diseases
Brief Title: Safety and Immunogenicity of Adjuvanted SARS-CoV-2 (SCB-2019) Vaccine in Adults With Chronic Immune-Mediated Diseases
Acronym: COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was early terminated considering the inability to enroll the required study population.
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-005
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hepatitis A Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCB-2019 Group (Experimental): CpG 1018/Alum-adjuvanted SCB-2019 vaccine
  Interventions: Biological: CpG 1018/Alum-adjuvanted SCB-2019 vaccine
- Control Group (Placebo Comparator): Havrix and Placebo
  Interventions: Biological: Havrix; Other: Placebo; 0.9% saline

INTERVENTIONS:
Biological: CpG 1018/Alum-adjuvanted SCB-2019 vaccine — Participants will receive 1 intramuscular (IM) injection of 30 microgram (mcg) SCB-2019 with CpG 1018/Alum adjuvant on Day 1 and on Day 22.
  Arms: SCB-2019 Group
Biological: Havrix — Participants will receive Havrix (Hepatitis A vaccine) containing 1440 Enzyme-linked Immunosorbent Assay (ELISA) units (EL.U.) in 1.0 mL dose on Day 1.
  Other Names: Hepatitis A vaccine
  Arms: Control Group
Other: Placebo; 0.9% saline — Participants will receive 1 IM injection of SCB-2019-matching placebo on Day 22.
  Arms: Control Group

SUMMARY:
The purpose of the study is to evaluate the safety and immunogenicity of the investigational CpG 1018/Alum-adjuvanted recombinant SARS-CoV-2 trimeric spike (S)-protein subunit vaccine (SCB-2019) in adult participants with stable chronic inflammatory immune-mediated diseases (IMDs), compared to control vaccine.

DETAILED DESCRIPTION:
This study is to evaluate the safety and immunogenicity of the investigational CpG 1018/Alum-adjuvanted recombinant SARS-CoV-2 trimeric S-protein subunit vaccine (SCB 2019) compared with control. Approximately 300 study participants with rheumatoid arthritis (RA), inflammatory bowel disease (IBD) and relapsing-remitting multiple sclerosis (RRMS) will be randomized according a 1:1 ratio to receive SCB-2019 or control vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female greater than or equal to (>=) 18 years of age.
2. Participants who are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.
3. Participants are willing and able to give an informed consent, prior to screening.
4. Participants should be in generally good health except for the following chronic immune-mediated diseases:

   * RA who received chronic ([>=] 3 months) immunosuppressive therapy with immunomodulators (such as methotrexate and abatacept), TNF-alpha inhibitors (such as etanercept, adalimumab, certolizumab, golimumab or infliximab), janus kinase (JAK) Inhibitors (such as tofacitinib or baricitinib), or Interleukin-6 (IL-6) receptor inhibitors (such as tocilizumab).
   * IBD: (Crohn's disease, Ulcerative colitis or Indeterminate colitis) who received chronic ([>=] 3 months) immunosuppressive therapy with TNF-alpha inhibitors (such as infliximab or adalimumab), immunomodulators (such as 6- mercaptopurine, azathioprine, or methotrexate), corticosteroids (such as prednisone, prednisolone, or methylprednisolone), or tacrolimus.
   * RRMS who received chronic ([>=] 6 months) stable disease modifying therapy (DMT) with platform therapeutics (beta-interferons, glatirameracetate, teriflunomide, dimethylfumarate), Sphingosine-1-phosphate receptor (S1PR) modulators (fingolimod, ozanimod, siponimod) or monoclonals (natalizumab).
5. Participants should be in remission (RA, IBD), or have low disease activity (RA) or stable disease (RRMS) without modification of immunosuppressive therapy (i.e. no dose change, no medication change, no rescue therapy) for at least 3 months (6 months for RRMS) prior to enrollment and not anticipated to undergo a change in immunosuppressive therapy for 1 month after Dose 2.
6. Female participant are eligible to participate in the study if not pregnant and breastfeeding.
7. Male participants must agree to employ acceptable contraception from the day of first dose of the study vaccine and during the entire study period and also refrain from donating sperm during this period.

Exclusion Criteria:

1. Participants with fever > 37.5°C (irrespective of method), or any acute illness at baseline (Day 1) or within 3 days prior to randomization. Participants meeting this criterion may be rescheduled (within the relevant window). Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
2. Participants with confirmed SARS-CoV-2 infection (as defined by Rapid COVID Antigen Test or an equivalent at Visit 1) or with history of COVID-19.
3. Participants who have received a prior investigational or licensed COVID-19 vaccine, or previous hepatitis A vaccine 12 months prior to Day 1.
4. Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, HIV infection) or having received systemic corticosteroids and/or immunosuppressive/cytotoxic therapy (e.g., medications used for cancer chemotherapy, organ transplantation or to treat autoimmune disorders other than RA, IBD or RRMS) within 6 months prior to enrollment.
5. Participants with any progressive unstable or uncontrolled clinical conditions.
6. Participants with surgery scheduled during the study period.
7. Participants who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccines, such as hepatitis A vaccine (as outlined in the Havrix Summary of Product Characteristics, EU SmPC, GSK, 2020), or CpG 1018/Alum/SCB-2019 components as outlined in the latest IB.
8. Participants who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
9. Participants who have received any other investigational product within 3 months to Day 1 or intent to participate in another clinical study at any time during the conduct of this study.
10. Participants who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 14 days after the second vaccination.
11. Participants with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection.
12. Participants who have received treatment with Rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to enrollment or planned during the study period.
13. Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period.
14. Participants with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional participant risk.
15. Participants with any seizure disorder, or history of Guillian-Barré syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Unsolicited Adverse Events (AEs) | Day 1 through Day 43
Percentage of Participants With Medically Attended AEs (MAAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | Day 1 through Day 205
Percentage of Participants With Any Confirmed Relapse of Immune-mediated Disease (RA, IBD, or RRMS) | Day 1 through Day 205

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) in Participants With RA, IBD, and RRMS | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb in Participants With RA, IBD, and RRMS | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb in Participants With RA, IBD and RRMS | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody in Participants With RA, IBD, and RRMS | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody in Participants With RA, IBD, and RRMS | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody in Participants With RA, IBD, and RRMS | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) in Participants Who Receive Corticosteroids | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb in Participants Who Receive Corticosteroids | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb in Participants Who Receive Corticosteroids | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody in Participants Who Receive Corticosteroids | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody in Participants Who Receive Corticosteroids | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody in Participants Who Receive Corticosteroids | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) in Participants Who Receive Tumor Necrosis Factor (TNF)-alpha Inhibitors | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb in Participants Who Receive TNF-alpha Inhibitors | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb in Participants who Received TNF-alpha Inhibitors | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody in Participants Who Receive TNF-alpha Inhibitors | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody in Participants Who Receive TNF-alpha Inhibitors | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody in Participants Who Receive TNF-alpha Inhibitors | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) in Participants Who Receive Immunomodulators | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb in Participants Who Receive Immunomodulators | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb in Participants who Receive Immunomodulators | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody in Participants Who Receive Immunomodulators | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody in Participants Who Receive Immunomodulators | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody in Participants Who Receive Immunomodulators | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody (nAb) in Participants Who Receive Other Treatment Regimens | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb in Participants Who Receive Other Treatment Regimens | Day 22, 36 and 205
Number of Participants With Seroconversion for SARS-CoV-2 nAb in Participants Who Receive Other Treatment Regimens | Day 22, 36 and 205
Geometric Mean Titer (GMT) of SCB-2019 Binding Antibody in Participants Who Receive Other Treatment Regimens | Day 1, 22, 36 and 205
Geometric Mean Fold Rise (GMFRs) of SCB-2019 Binding Antibody in Participants Who Receive Other Treatment Regimens | Day 22, 36 and 205
Number of Participants With Seroconversion for SCB-2019 Binding Antibody in Participants Who Receive Other Treatment Regimens | Day 22, 36 and 205
Number of Participants With Local and Systemic Solicited AEs | Day 1 to 7 and Day 22 to 29

CONTACTS AND LOCATIONS:
Locations (4):
- Ukraine (4):
  - Medical Centre of Edelweiss Medics LLC, Kyiv
  - Medical Center of Medbud-Clinic LLC, Kyiv
  - Center of Family Medicine Plus, LLC, Kyiv
  - Medical Center Salutem LLC, Vinnitsa